CLINICAL TRIAL: NCT03219398
Title: Comparison Effect Between Lower Pressure and Standard Pressure Pneumoperitoneum on Sign of Acute Systemic Inflammation, Endothelial Injury, and Acute Kidney Injury: A Randomized Clinical Trial in Living Donor Laparoscopic Nephrectomy
Brief Title: The Effect of Lower Intraabdominal Pressure on Syndecan-1, sVEGF-R2, Occludin, KIM-1, and IL-6 on Living Donor Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Anesthesiologist Consultant, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes020
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Living donor laparoscopic nephrectomy; Pneumoperitoneum; Renal resistive index; Syndecan-1; soluble VEGF-R2; Occludin; KIM-1; Interleukin-6
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-10 mmHg (Active Comparator): Patients receive lower pneumoperitoneum pressure
  Interventions: Procedure: Pneumoperitoneum pressure
- 12-14 mmHg (Active Comparator): Patients receive higher pneumoperitoneum pressure
  Interventions: Procedure: Pneumoperitoneum pressure

INTERVENTIONS:
Procedure: Pneumoperitoneum pressure — Subjects were set to 8- 10 mmHg pressure during laparoscopic surgery; Subjects were set to 12-14 mmHg pressure during laparoscopic surgery

SUMMARY:
This study aimed to evaluate the increase of intraabdominal pressure 12- 14 mmHg caused by pneumoperitoneum resulted from carbon dioxide (CO2) insufflation induce glycocalyx endothelial injury that cause kidney tubular injury on live donor patient that undergo laparoscopic nephrectomy surgery, and decreasing the intraabdominal pressure to 8-10 mmHg during surgery is expected to reduce the injury.

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups. Intravenous (IV) cannula (18-20G) with Ringer Lactate fluid, non-invasive blood pressure monitor, electrocardiogram (ECG), ICON® monitor, hemodynamic monitor and pulse-oxymetry were set on the subjects in the operation room. Premedication with 2 mg IV midazolam and 1 mcg/kg IV fentanyl as premedication. General anesthesia induction was done by fentanyl 4 mcg/kg, propofol 1-2 mg/kg, and rocuronium 0,5 mg/kg. Maintenance was done by sevoflurane 1 minimum alveolar concentration (MAC), fentanyl and rocuronium with bupivacaine bolus 6ml every 90 minutes. Surgery starts with patient in lumbotomy position laterally, CO2 gas insufflated during the installment of laparoscopy probe until it reaches 10- 12 mmHg pressure. Laparoscopy targeted the pneumoperitoneum pressure until 8- 10 mmHg or 12- 14 mmHg depends on subject randomization. Surgery duration, blood pressure, heart rate, respiratory rate, oxygen saturation (SpO2) were recorded. During surgery, blood sample for interleukin (IL)-6, Syndecan-1, sVGEF-R2, Occludin and KIM-1 urine were taken before the anesthesia induction as the baseline; 2 hours of gas insufflation intraoperatively; and 2 hours after gas desufflation. The measurement of renal artery and kidney lobe artery that undergo nephrectomy, will be measured by convex probe 3.5-5 megahertz (MHz) ultrasonography (USG) Logic 7-GE or Sonosite. The measurement of RI was done on the left kidney at the time: before the anesthesia induction as the baseline; 2 hours of gas insufflation intraoperatively; and 2 hours after gas desufflation on the remaining right kidney. All patients received bilateral Quadratus Lumborum (QL) block using bupivacaine 0.25% before extubation. Patient were extubated until fully conscious and can follow command verbally. Patient will be transported in recovery room post operation. Data was analyzed using SPSS (Statistical Package for Social Scientist), for parametric unpaired data is using unpaired T-test or One way ANOVA test, ffor unpaired non parametric data using Mann Whitney or Kruskal-Wallis. Non Parametric continuous data using Wilcoxon's signed rank test or Friedman Test. Categorical data using Chi-square. For numerical data more than 1 measurement will be analysed using Comparative General Linear Model. Data normality was tested by Kolmogorov-Smirnov test. Significant value is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-60 years old undergoing laparoscopic surgery, with American Society of Anesthesiologist (ASA) 1, body mass index 18-25. Patients who agreed to participate in this study and sign informed consent.

Exclusion Criteria:

* Subjects in the outside criteria of American Society of Anesthesia 1, body mass index >25.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in Syndecan-1 level from baseline | 24 hours
  Measurement of plasma Syndecan-1 level after patient is sedated at baseline, 2 hours insufflation, and 2 hours after desufflation
Changes in sVGEFR-2 level from baseline | 24 hours
  Measurement of plasma soluble VGEF-R2 level after patient is sedated at baseline, 2 hours insufflation, and 2 hours after desufflation
Changes in KIM-1 level from baseline | 24 hours
  Measurement of Urinary KIM-1 level after patient is sedated at baseline, 2 hours insufflation, and 2 hours after desufflation
Changes in Interleukin-6 from baseline | 24 hours
  Measurement of plasma Interleukin-6 after patient is sedated at baseline, 2 hours insufflation, and 2 hours after desufflation

SECONDARY OUTCOMES:
Changes in Renal Resistive Index from baseline | 24 hours
  Measurement of Renal artery resistive index using ultrasound after patient is sedated at baseline, 2 hours insufflation, and 2 hours after desufflation
Renal biopsy tissue Syndecan-1 | 24 hours
  Histopathology and immunostaining Syndecan-1 of renal biopsy after donor kidney has been removed from patient and stored in ice
Intraoperative fentanyl dosage | 24 hours
  Comparison of fentanyl needs during operation
Changes in Occludin level from baseline | 24 hours
  Measurement of plasma Occludin level after patient is sedated at baseline, 2 hours insufflation, and 2 hours after desufflation

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, MD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fehrman-Ekholm I, Lennerling A, Kvarnstrom N, Rizell M, Olausson M. [Living donor kidney transplantation--a successful story. Very cost-effective--and the donors live long with good health]. Lakartidningen. 2011 Nov 30-Dec 6;108(48):2492-5. No abstract available. Swedish. PMID 22462270
- [Background] Choi JD, Park JW, Choi JY, Kim HS, Jeong BC, Jeon SS, Lee HM, Choi HY, Seo SI. Renal damage caused by warm ischaemia during laparoscopic and robot-assisted partial nephrectomy: an assessment using Tc 99m-DTPA glomerular filtration rate. Eur Urol. 2010 Dec;58(6):900-5. doi: 10.1016/j.eururo.2010.08.044. Epub 2010 Sep 15. PMID 21414862
- [Background] Vasdev N, Poon AS, Gowrie-Mohan S, Lane T, Boustead G, Hanbury D, Adshead JM. The physiologic and anesthetic considerations in elderly patients undergoing robotic renal surgery. Rev Urol. 2014;16(1):1-9. PMID 24791150
- [Background] Dalfino L, Tullo L, Donadio I, Malcangi V, Brienza N. Intra-abdominal hypertension and acute renal failure in critically ill patients. Intensive Care Med. 2008 Apr;34(4):707-13. doi: 10.1007/s00134-007-0969-4. Epub 2007 Dec 19. PMID 18157662
- [Background] Mohmand H, Goldfarb S. Renal dysfunction associated with intra-abdominal hypertension and the abdominal compartment syndrome. J Am Soc Nephrol. 2011 Apr;22(4):615-21. doi: 10.1681/ASN.2010121222. Epub 2011 Feb 10. PMID 21310818
- [Background] Nguyen NT, Perez RV, Fleming N, Rivers R, Wolfe BM. Effect of prolonged pneumoperitoneum on intraoperative urine output during laparoscopic gastric bypass. J Am Coll Surg. 2002 Oct;195(4):476-83. doi: 10.1016/s1072-7515(02)01321-2. PMID 12375752
- [Background] Garg AX, Muirhead N, Knoll G, Yang RC, Prasad GV, Thiessen-Philbrook H, Rosas-Arellano MP, Housawi A, Boudville N; Donor Nephrectomy Outcomes Research (DONOR) Network. Proteinuria and reduced kidney function in living kidney donors: A systematic review, meta-analysis, and meta-regression. Kidney Int. 2006 Nov;70(10):1801-10. doi: 10.1038/sj.ki.5001819. Epub 2006 Sep 27. PMID 17003822
- [Background] Gomez-Anson B, Carrero-Lopez V, Diaz-Gonzalez R. Image-directed color Doppler ultrasound evaluation of the single kidney after unilateral nephrectomy in adults. J Clin Ultrasound. 1997 Jan;25(1):29-35. doi: 10.1002/(sici)1097-0096(199701)25:13.0.co;2-m. PMID 9010805
- [Background] Nekouei S, Ahmadnia H, Abedi M, Alamolhodaee MH, Abedi MS. Resistive index of the remaining kidney in allograft kidney donors. Exp Clin Transplant. 2012 Oct;10(5):454-7. doi: 10.6002/ect.2012.0054. PMID 23031084
- [Background] Lindberg F, Bergqvist D, Bjorck M, Rasmussen I. Renal hemodynamics during carbon dioxide pneumoperitoneum: an experimental study in pigs. Surg Endosc. 2003 Mar;17(3):480-4. doi: 10.1007/s00464-002-9044-y. Epub 2002 Nov 6. PMID 12415336
- [Background] Wiesenthal JD, Fazio LM, Perks AE, Blew BD, Mazer D, Hare G, Honey RJ, Pace KT. Effect of pneumoperitoneum on renal tissue oxygenation and blood flow in a rat model. Urology. 2011 Jun;77(6):1508.e9-15. doi: 10.1016/j.urology.2011.02.022. Epub 2011 Apr 19. PMID 21507469
- [Background] Zacherl J, Thein E, Stangl M, Feussner H, Bock S, Mittlbock M, Erhardt W, Siewert JR. The influence of periarterial papaverine application on intraoperative renal function and blood flow during laparoscopic donor nephrectomy in a pig model. Surg Endosc. 2003 Aug;17(8):1231-6. doi: 10.1007/s00464-002-8835-5. Epub 2003 Jun 13. PMID 12799887
- [Background] Gudmundsson FF, Viste A, Myking OL, Bostad L, Grong K, Svanes K. Role of angiotensin II under prolonged increased intraabdominal pressure (IAP) in pigs. Surg Endosc. 2003 Jul;17(7):1092-7. doi: 10.1007/s00464-002-9123-0. Epub 2003 Mar 14. PMID 12632126
- [Background] Borba MR, Lopes RI, Carmona M, Neto BM, Nahas SC, Pereira PR. Effects of enalaprilat on the renin-angiotensin-aldosterone system and on renal function during CO2 pneumoperitoneum. J Endourol. 2005 Oct;19(8):1026-31. doi: 10.1089/end.2005.19.1026. PMID 16253075
- [Background] Demyttenaere S, Feldman LS, Fried GM. Effect of pneumoperitoneum on renal perfusion and function: a systematic review. Surg Endosc. 2007 Feb;21(2):152-60. doi: 10.1007/s00464-006-0250-x. Epub 2006 Dec 9. PMID 17160650
- [Background] Warle MC, Berkers AW, Langenhuijsen JF, van der Jagt MF, Dooper PM, Kloke HJ, Pilzecker D, Renes SH, Wever KE, Hoitsma AJ, van der Vliet JA, D'Ancona FC. Low-pressure pneumoperitoneum during laparoscopic donor nephrectomy to optimize live donors' comfort. Clin Transplant. 2013 Jul-Aug;27(4):E478-83. doi: 10.1111/ctr.12143. Epub 2013 Jun 24. PMID 23795745
- [Background] Lindstrom P, Wadstrom J, Ollerstam A, Johnsson C, Persson AE. Effects of increased intra-abdominal pressure and volume expansion on renal function in the rat. Nephrol Dial Transplant. 2003 Nov;18(11):2269-77. doi: 10.1093/ndt/gfg362. PMID 14551353
- [Background] Cisek LJ, Gobet RM, Peters CA. Pneumoperitoneum produces reversible renal dysfunction in animals with normal and chronically reduced renal function. J Endourol. 1998 Apr;12(2):95-100. doi: 10.1089/end.1998.12.95. PMID 9607433
- [Background] Carmona M, Lopes RI, Borba M, Omokawa M, Naufal R, Miyaji K, Matsumura N, Vieira N, Pereira PR. Comparison of the effects of carbon dioxide and helium pneumoperitoneum on renal function. J Endourol. 2008 May;22(5):1077-82. doi: 10.1089/end.2007.0369. PMID 18419332
- [Background] Sammour T, Mittal A, Loveday BP, Kahokehr A, Phillips AR, Windsor JA, Hill AG. Systematic review of oxidative stress associated with pneumoperitoneum. Br J Surg. 2009 Aug;96(8):836-50. doi: 10.1002/bjs.6651. PMID 19591166
- [Background] Yilmaz S, Koken T, Tokyol C, Kahraman A, Akbulut G, Serteser M, Polat C, Gokce C, Gokce O. Can preconditioning reduce laparoscopy-induced tissue injury? Surg Endosc. 2003 May;17(5):819-24. doi: 10.1007/s00464-002-9096-z. Epub 2003 Jan 18. PMID 12584602
- [Background] Golab F, Kadkhodaee M, Zahmatkesh M, Hedayati M, Arab H, Schuster R, Zahedi K, Lentsch AB, Soleimani M. Ischemic and non-ischemic acute kidney injury cause hepatic damage. Kidney Int. 2009 Apr;75(8):783-92. doi: 10.1038/ki.2008.683. Epub 2009 Jan 28. PMID 19177157
- [Background] Yap S, Park SW, Egan B, Lee HT. Cytokine elevation and transaminitis after laparoscopic donor nephrectomy. Am J Physiol Renal Physiol. 2012 May 1;302(9):F1104-11. doi: 10.1152/ajprenal.00543.2011. Epub 2012 Jan 18. PMID 22262478
- [Background] Khoury W, Jakowlev K, Fein A, Orenstein H, Nakache R, Weinbroum AA. Renal apoptosis following carbon dioxide pneumoperitoneum in a rat model. J Urol. 2008 Oct;180(4):1554-8. doi: 10.1016/j.juro.2008.06.008. Epub 2008 Aug 16. PMID 18710725
- [Background] Seguro AC, Poli de Figueiredo LF, Shimizu MH. N-acetylcysteine (NAC) protects against acute kidney injury (AKI) following prolonged pneumoperitoneum in the rat. J Surg Res. 2012 Jun 15;175(2):312-5. doi: 10.1016/j.jss.2011.05.052. Epub 2011 Jun 23. PMID 21764077
- [Background] Matsuzaki S, Botchorishvili R, Jardon K, Maleysson E, Canis M, Mage G. Impact of intraperitoneal pressure and duration of surgery on levels of tissue plasminogen activator and plasminogen activator inhibitor-1 mRNA in peritoneal tissues during laparoscopic surgery. Hum Reprod. 2011 May;26(5):1073-81. doi: 10.1093/humrep/der055. Epub 2011 Mar 9. PMID 21393301
- [Background] De Souza D, Costa WS, Cardoso LEM, Benchimol M, Pereira-Sampaio MA, Sampaio FJB. Prolonged pneumoperitoneum did not harm the kidney in a rat model. J Urol 2012;187(4):412-3.
- [Background] Arsalani-Zadeh R, Ullah S, Khan S, MacFie J. Oxidative stress in laparoscopic versus open abdominal surgery: a systematic review. J Surg Res. 2011 Jul;169(1):e59-68. doi: 10.1016/j.jss.2011.01.038. Epub 2011 Feb 22. PMID 21492871
- [Background] Hoogendijk-van den Akker JM, Warle MC, van Zuilen AD, Kloke HJ, Wever KE, d'Ancona FC, Ӧzdemir DM, Wetzels JF, Hoitsma AJ. Urinary biomarkers after donor nephrectomy. Transpl Int. 2015 May;28(5):544-52. doi: 10.1111/tri.12523. Epub 2015 Feb 2. PMID 25581388
- [Background] Mishra J, Ma Q, Prada A, Mitsnefes M, Zahedi K, Yang J, Barasch J, Devarajan P. Identification of neutrophil gelatinase-associated lipocalin as a novel early urinary biomarker for ischemic renal injury. J Am Soc Nephrol. 2003 Oct;14(10):2534-43. doi: 10.1097/01.asn.0000088027.54400.c6. PMID 14514731
- [Background] Ballinger ML, Nigro J, Frontanilla KV, Dart AM, Little PJ. Regulation of glycosaminoglycan structure and atherogenesis. Cell Mol Life Sci. 2004 Jun;61(11):1296-306. doi: 10.1007/s00018-004-3389-4. PMID 15170508
- [Background] Smit M, Hofker HS, Leuvenink HG, Krikke C, Jongman RM, Zijlstra JG, van Meurs M. A human model of intra-abdominal hypertension: even slightly elevated pressures lead to increased acute systemic inflammation and signs of acute kidney injury. Crit Care. 2013 Apr 4;17(2):425. doi: 10.1186/cc12568. No abstract available. PMID 23566574
- [Background] Malbrain ML, Vidts W, Ravyts M, De Laet I, De Waele J. Acute intestinal distress syndrome: the importance of intra-abdominal pressure. Minerva Anestesiol. 2008 Nov;74(11):657-73. Epub 2008 Apr 18. PMID 18636062
- [Background] United States Renal Data System. USRDS 2013 annual data report: atlas of chronic kidney disease and end-stage re- nal disease in the United States. Bethesda, MD: National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, 2013.
- [Background] Department of Health and Human Services, Health Resources and Services Administration. Organ Procurement and Transplantation Network. Available from URL: http:// optn.transplant.hrsa.gov/converge/latest- Data/rptData.asp.
- [Background] Harjito FV. One-Year Survival of Kidney Transplant Recipients in Cipto Mangunkusumo Hospital. Perpustakaan Fakultas Kedokteran Universitas Indonesia 2015. Available from URL: http://perpustakaan.fk.ui.ac.id/opac/index.resipien+transplantasi+ginjal.
- [Background] Yang SL, Harkaway R, Badosa F, Ginsberg P, Greenstein MA. Minimal incision living donor nephrectomy: improvement in patient outcome. Urology. 2002 May;59(5):673-7. doi: 10.1016/s0090-4295(02)01516-9. PMID 11992838
- [Background] Ratner LE, Ciseck LJ, Moore RG, Cigarroa FG, Kaufman HS, Kavoussi LR. Laparoscopic live donor nephrectomy. Transplantation. 1995 Nov 15;60(9):1047-9. PMID 7491680
- [Background] Nogueira JM, Cangro CB, Fink JC, Schweitzer E, Wiland A, Klassen DK, Gardner J, Flowers J, Jacobs S, Cho E, Philosophe B, Bartlett ST, Weir MR. A comparison of recipient renal outcomes with laparoscopic versus open live donor nephrectomy. Transplantation. 1999 Mar 15;67(5):722-8. doi: 10.1097/00007890-199903150-00014. PMID 10096529
- [Background] Barth RN. Donor Nephrectomy. Kidney Transplantation Principle 2013;8:118-29.
- [Background] Vats HS, Rayhill SC, Thomas CP. Early postnephrectomy donor renal function: laparoscopic versus open procedure. Transplantation. 2005 Mar 15;79(5):609-12. doi: 10.1097/01.tp.0000151662.84962.4e. PMID 15753853
- [Background] Binda MM. Humidification during laparoscopic surgery: overview of the clinical benefits of using humidified gas during laparoscopic surgery. Arch Gynecol Obstet. 2015 Nov;292(5):955-71. doi: 10.1007/s00404-015-3717-y. Epub 2015 Apr 25. PMID 25911545
- [Background] Koivusalo AM, Kellokumpu I, Scheinin M, Tikkanen I, Halme L, Lindgren L. Randomized comparison of the neuroendocrine response to laparoscopic cholecystectomy using either conventional or abdominal wall lift techniques. Br J Surg. 1996 Nov;83(11):1532-6. doi: 10.1002/bjs.1800831112. PMID 9014667
- [Background] Joris JL, Noirot DP, Legrand MJ, Jacquet NJ, Lamy ML. Hemodynamic changes during laparoscopic cholecystectomy. Anesth Analg. 1993 May;76(5):1067-71. doi: 10.1213/00000539-199305000-00027. PMID 8484509
- [Background] Gutt CN, Kim ZG, Schemmer P, Krahenbuhl L, Schmedt CG. Impact of laparoscopic and conventional surgery on Kupffer cells, tumor-associated CD44 expression, and intrahepatic tumor spread. Arch Surg. 2002 Dec;137(12):1408-12. doi: 10.1001/archsurg.137.12.1408. PMID 12470109
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Hazebroek EJ, de Vos tot Nederveen Cappel R, Gommers D, van Gelder T, Weimar W, Steyerberg EW, Bonjer HJ, IJzermans JN. Antidiuretic hormone release during laparoscopic donor nephrectomy. Arch Surg. 2002 May;137(5):600-4; discussion 605. doi: 10.1001/archsurg.137.5.600. PMID 11982475
- [Background] Kehlet H. Surgical stress response: does endoscopic surgery confer an advantage? World J Surg. 1999 Aug;23(8):801-7. doi: 10.1007/s002689900583. PMID 10415206
- [Background] Donald RA, Perry EG, Wittert GA, Chapman M, Livesey JH, Ellis MJ, Evans MJ, Yandle T, Espiner EA. The plasma ACTH, AVP, CRH and catecholamine responses to conventional and laparoscopic cholecystectomy. Clin Endocrinol (Oxf). 1993 Jun;38(6):609-15. doi: 10.1111/j.1365-2265.1993.tb02142.x. PMID 8392916
- [Background] Altintas F, Tunali Y, Bozkurt P, Kaya G, Uygun N, Aricioglu F, Hacibekiroglu M. An experimental study on the relationship of intra-abdominal pressure and renal ischemia. Middle East J Anaesthesiol. 2001 Feb;16(1):55-66. PMID 11281048
- [Background] Mikami O, Kawakita S, Fujise K, Shingu K, Takahashi H, Matsuda T. Catecholamine release caused by carbon dioxide insufflation during laparoscopic surgery. J Urol. 1996 Apr;155(4):1368-71. PMID 8632576
- [Background] Siniscalchi A, Gamberini L, Laici C, Bardi T, Faenza S. Thoracic epidural anesthesia: Effects on splanchnic circulation and implications in Anesthesia and Intensive care. World J Crit Care Med. 2015 Feb 4;4(1):89-104. doi: 10.5492/wjccm.v4.i1.89. eCollection 2015 Feb 4. PMID 25685727
- [Background] Janssen-Heininger YM, Mossman BT, Heintz NH, Forman HJ, Kalyanaraman B, Finkel T, Stamler JS, Rhee SG, van der Vliet A. Redox-based regulation of signal transduction: principles, pitfalls, and promises. Free Radic Biol Med. 2008 Jul 1;45(1):1-17. doi: 10.1016/j.freeradbiomed.2008.03.011. Epub 2008 Mar 27. PMID 18423411
- [Background] Whelan RL, Franklin M, Holubar SD, Donahue J, Fowler R, Munger C, Doorman J, Balli JE, Glass J, Gonzalez JJ, Bessler M, Xie H, Treat M. Postoperative cell mediated immune response is better preserved after laparoscopic vs open colorectal resection in humans. Surg Endosc. 2003 Jun;17(6):972-8. doi: 10.1007/s00464-001-8263-y. Epub 2003 Mar 19. PMID 12640542
- [Background] Del Rio D, Stewart AJ, Pellegrini N. A review of recent studies on malondialdehyde as toxic molecule and biological marker of oxidative stress. Nutr Metab Cardiovasc Dis. 2005 Aug;15(4):316-28. doi: 10.1016/j.numecd.2005.05.003. PMID 16054557
- [Background] Comporti M, Signorini C, Arezzini B, Vecchio D, Monaco B, Gardi C. F2-isoprostanes are not just markers of oxidative stress. Free Radic Biol Med. 2008 Feb 1;44(3):247-56. doi: 10.1016/j.freeradbiomed.2007.10.004. Epub 2007 Oct 13. PMID 17997380
- [Background] Betteridge DJ. What is oxidative stress? Metabolism. 2000 Feb;49(2 Suppl 1):3-8. doi: 10.1016/s0026-0495(00)80077-3. PMID 10693912
- [Background] Akbulut G, Polat C, Aktepe F, Yilmaz S, Kahraman A, Serteser M, Gokce C, Gokce O. The oxidative effect of prolonged CO2 pneumoperitoneum on renal tissue of rats. Surg Endosc. 2004 Sep;18(9):1384-8. doi: 10.1007/s00464-003-9114-9. Epub 2004 Jun 29. PMID 15803240
- [Background] Akbulut G, Serteser M, Polat C, Koken T, Aktepe F, Yilmaz S, Gokce C, Gokce O. Changes in tissue-oxidative stress markers in an experimental model of laparoscopic donor nephrectomy. Transplantation. 2002 Dec 27;74(12):1768-72. doi: 10.1097/01.TP.0000038730.30170.24. PMID 12499896
- [Background] Demirbas M, Samli M, Aksoy Y, Guler C, Kilinc A, Dincel C. Comparison of changes in tissue oxidative-stress markers in experimental model of open, laparoscopic, and retroperitoneoscopic donor nephrectomy. J Endourol. 2004 Feb;18(1):105-8. doi: 10.1089/089277904322836758. PMID 15006062
- [Background] Diebel LN, Dulchavsky SA, Wilson RF. Effect of increased intra-abdominal pressure on mesenteric arterial and intestinal mucosal blood flow. J Trauma. 1992 Jul;33(1):45-8; discussion 48-9. doi: 10.1097/00005373-199207000-00010. PMID 1635105
- [Background] Pross M, Schulz HU, Flechsig A, Manger T, Halangk W, Augustin W, Lippert H, Reinheckel T. Oxidative stress in lung tissue induced by CO(2) pneumoperitoneum in the rat. Surg Endosc. 2000 Dec;14(12):1180-4. doi: 10.1007/s004640000189. PMID 11148794
- [Background] Bentes de Souza AM, Rogers MS, Wang CC, Yuen PM, Ng PS. Comparison of peritoneal oxidative stress during laparoscopy and laparotomy. J Am Assoc Gynecol Laparosc. 2003 Feb;10(1):65-74. doi: 10.1016/s1074-3804(05)60237-x. PMID 12554997
- [Background] Zulfikaroglu B, Koc M, Soran A, Isman FK, Cinel I. Evaluation of oxidative stress in laparoscopic cholecystectomy. Surg Today. 2002;32(10):869-74. doi: 10.1007/s005950200169. PMID 12376782
- [Background] Veskoukis AS, Nikolaidis MG, Kyparos A, Kouretas D. Blood reflects tissue oxidative stress depending on biomarker and tissue studied. Free Radic Biol Med. 2009 Nov 15;47(10):1371-4. doi: 10.1016/j.freeradbiomed.2009.07.014. Epub 2009 Jul 17. PMID 19616614
- [Background] Ozmen MM, Kessaf Aslar A, Besler HT, Cinel I. Does splanchnic ischemia occur during laparoscopic cholecystectomy? Surg Endosc. 2002 Mar;16(3):468-71. doi: 10.1007/s00464-001-9031-8. Epub 2001 Nov 16. PMID 11928030
- [Background] Sare M, Hamamci D, Yilmaz I, Birincioglu M, Mentes BB, Ozmen M, Yesilada O. Effects of carbon dioxide pneumoperitoneum on free radical formation in lung and liver tissues. Surg Endosc. 2002 Jan;16(1):188-92. doi: 10.1007/s004640090103. Epub 2001 Oct 5. PMID 11961637
- [Background] Windberger UB, Auer R, Keplinger F, Langle F, Heinze G, Schindl M, Losert UM. The role of intra-abdominal pressure on splanchnic and pulmonary hemodynamic and metabolic changes during carbon dioxide pneumoperitoneum. Gastrointest Endosc. 1999 Jan;49(1):84-91. doi: 10.1016/s0016-5107(99)70450-5. PMID 9869728
- [Background] Ishizaki Y, Bandai Y, Shimomura K, Abe H, Ohtomo Y, Idezuki Y. Safe intraabdominal pressure of carbon dioxide pneumoperitoneum during laparoscopic surgery. Surgery. 1993 Sep;114(3):549-54. PMID 8367810
- [Background] Schilling MK, Redaelli C, Krahenbuhl L, Signer C, Buchler MW. Splanchnic microcirculatory changes during CO2 laparoscopy. J Am Coll Surg. 1997 Apr;184(4):378-82. PMID 9100683
- [Background] Polat C, Yilmaz S, Serteser M, Koken T, Kahraman A, Dilek ON. The effect of different intraabdominal pressures on lipid peroxidation and protein oxidation status during laparoscopic cholecystectomy. Surg Endosc. 2003 Nov;17(11):1719-22. doi: 10.1007/s00464-002-9258-z. Epub 2003 Sep 10. PMID 12958684
- [Background] Reitsma S, Slaaf DW, Vink H, van Zandvoort MA, oude Egbrink MG. The endothelial glycocalyx: composition, functions, and visualization. Pflugers Arch. 2007 Jun;454(3):345-59. doi: 10.1007/s00424-007-0212-8. Epub 2007 Jan 26. PMID 17256154
- [Background] Mulivor AW, Lipowsky HH. Inflammation- and ischemia-induced shedding of venular glycocalyx. Am J Physiol Heart Circ Physiol. 2004 May;286(5):H1672-80. doi: 10.1152/ajpheart.00832.2003. Epub 2004 Jan 2. PMID 14704229
- [Background] Sugahara K, Mikami T, Uyama T, Mizuguchi S, Nomura K, Kitagawa H. Recent advances in the structural biology of chondroitin sulfate and dermatan sulfate. Curr Opin Struct Biol. 2003 Oct;13(5):612-20. doi: 10.1016/j.sbi.2003.09.011. PMID 14568617
- [Background] Tkachenko E, Rhodes JM, Simons M. Syndecans: new kids on the signaling block. Circ Res. 2005 Mar 18;96(5):488-500. doi: 10.1161/01.RES.0000159708.71142.c8. PMID 15774861
- [Background] Jung U, Ley K. Regulation of E-selectin, P-selectin, and intercellular adhesion molecule 1 expression in mouse cremaster muscle vasculature. Microcirculation. 1997 Jun;4(2):311-9. doi: 10.3109/10739689709146794. PMID 9219223
- [Background] Kansas GS, Saunders KB, Ley K, Zakrzewicz A, Gibson RM, Furie BC, Furie B, Tedder TF. A role for the epidermal growth factor-like domain of P-selectin in ligand recognition and cell adhesion. J Cell Biol. 1994 Feb;124(4):609-18. doi: 10.1083/jcb.124.4.609. PMID 7508943
- [Background] Ruegg C, Mariotti A. Vascular integrins: pleiotropic adhesion and signaling molecules in vascular homeostasis and angiogenesis. Cell Mol Life Sci. 2003 Jun;60(6):1135-57. doi: 10.1007/s00018-003-2297-3. PMID 12861381
- [Background] Xiong JP, Stehle T, Goodman SL, Arnaout MA. Integrins, cations and ligands: making the connection. J Thromb Haemost. 2003 Jul;1(7):1642-54. doi: 10.1046/j.1538-7836.2003.00277.x. PMID 12871301
- [Background] Muller AM, Hermanns MI, Cronen C, Kirkpatrick CJ. Comparative study of adhesion molecule expression in cultured human macro- and microvascular endothelial cells. Exp Mol Pathol. 2002 Dec;73(3):171-80. doi: 10.1006/exmp.2002.2446. PMID 12565792
- [Background] Huxley VH, Curry FE. Differential actions of albumin and plasma on capillary solute permeability. Am J Physiol. 1991 May;260(5 Pt 2):H1645-54. doi: 10.1152/ajpheart.1991.260.5.H1645. PMID 2035684
- [Background] Tarbell JM, Weinbaum S, Kamm RD. Cellular fluid mechanics and mechanotransduction. Ann Biomed Eng. 2005 Dec;33(12):1719-23. doi: 10.1007/s10439-005-8775-z. PMID 16389519
- [Background] van den Berg BM, Vink H, Spaan JA. The endothelial glycocalyx protects against myocardial edema. Circ Res. 2003 Apr 4;92(6):592-4. doi: 10.1161/01.RES.0000065917.53950.75. Epub 2003 Mar 13. PMID 12637366
- [Background] van Haaren PM, VanBavel E, Vink H, Spaan JA. Localization of the permeability barrier to solutes in isolated arteries by confocal microscopy. Am J Physiol Heart Circ Physiol. 2003 Dec;285(6):H2848-56. doi: 10.1152/ajpheart.00117.2003. Epub 2003 Aug 7. PMID 12907418
- [Background] Rehm M, Zahler S, Lotsch M, Welsch U, Conzen P, Jacob M, Becker BF. Endothelial glycocalyx as an additional barrier determining extravasation of 6% hydroxyethyl starch or 5% albumin solutions in the coronary vascular bed. Anesthesiology. 2004 May;100(5):1211-23. doi: 10.1097/00000542-200405000-00025. PMID 15114220
- [Background] Levick JR, Michel CC. Microvascular fluid exchange and the revised Starling principle. Cardiovasc Res. 2010 Jul 15;87(2):198-210. doi: 10.1093/cvr/cvq062. Epub 2010 Mar 3. PMID 20200043
- [Background] Patel KD, Nollert MU, McEver RP. P-selectin must extend a sufficient length from the plasma membrane to mediate rolling of neutrophils. J Cell Biol. 1995 Dec;131(6 Pt 2):1893-902. doi: 10.1083/jcb.131.6.1893. PMID 8557755
- [Background] Vink H, Constantinescu AA, Spaan JA. Oxidized lipoproteins degrade the endothelial surface layer : implications for platelet-endothelial cell adhesion. Circulation. 2000 Apr 4;101(13):1500-2. doi: 10.1161/01.cir.101.13.1500. PMID 10747340
- [Background] Khan F, Galarraga B, Belch JJ. The role of endothelial function and its assessment in rheumatoid arthritis. Nat Rev Rheumatol. 2010 May;6(5):253-61. doi: 10.1038/nrrheum.2010.44. Epub 2010 Mar 30. PMID 20351705
- [Background] Gouverneur M, Spaan JA, Pannekoek H, Fontijn RD, Vink H. Fluid shear stress stimulates incorporation of hyaluronan into endothelial cell glycocalyx. Am J Physiol Heart Circ Physiol. 2006 Jan;290(1):H458-2. doi: 10.1152/ajpheart.00592.2005. Epub 2005 Aug 26. PMID 16126814
- [Background] van den Berg BM, Spaan JA, Rolf TM, Vink H. Atherogenic region and diet diminish glycocalyx dimension and increase intima-to-media ratios at murine carotid artery bifurcation. Am J Physiol Heart Circ Physiol. 2006 Feb;290(2):H915-20. doi: 10.1152/ajpheart.00051.2005. Epub 2005 Sep 9. PMID 16155109
- [Background] Quinsey NS, Greedy AL, Bottomley SP, Whisstock JC, Pike RN. Antithrombin: in control of coagulation. Int J Biochem Cell Biol. 2004 Mar;36(3):386-9. doi: 10.1016/s1357-2725(03)00244-9. PMID 14687916
- [Background] Tovar AM, de Mattos DA, Stelling MP, Sarcinelli-Luz BS, Nazareth RA, Mourao PA. Dermatan sulfate is the predominant antithrombotic glycosaminoglycan in vessel walls: implications for a possible physiological function of heparin cofactor II. Biochim Biophys Acta. 2005 Apr 15;1740(1):45-53. doi: 10.1016/j.bbadis.2005.02.008. Epub 2005 Mar 11. PMID 15878740
- [Background] Weiler H, Isermann BH. Thrombomodulin. J Thromb Haemost. 2003 Jul;1(7):1515-24. doi: 10.1046/j.1538-7836.2003.00306.x. PMID 12871287
- [Background] Becker BF, Chappell D, Bruegger D, Annecke T, Jacob M. Therapeutic strategies targeting the endothelial glycocalyx: acute deficits, but great potential. Cardiovasc Res. 2010 Jul 15;87(2):300-10. doi: 10.1093/cvr/cvq137. Epub 2010 May 11. PMID 20462866
- [Background] Steppan J, Hofer S, Funke B, Brenner T, Henrich M, Martin E, Weitz J, Hofmann U, Weigand MA. Sepsis and major abdominal surgery lead to flaking of the endothelial glycocalix. J Surg Res. 2011 Jan;165(1):136-41. doi: 10.1016/j.jss.2009.04.034. Epub 2009 May 20. PMID 19560161
- [Background] Suwarto S, Sasmono RT, Sinto R, Ibrahim E, Suryamin M. Association of Endothelial Glycocalyx and Tight and Adherens Junctions With Severity of Plasma Leakage in Dengue Infection. J Infect Dis. 2017 Mar 15;215(6):992-999. doi: 10.1093/infdis/jix041. PMID 28453844
- [Background] Jeansson M, Haraldsson B. Morphological and functional evidence for an important role of the endothelial cell glycocalyx in the glomerular barrier. Am J Physiol Renal Physiol. 2006 Jan;290(1):F111-6. doi: 10.1152/ajprenal.00173.2005. Epub 2005 Aug 9. PMID 16091582
- [Background] Hayat MA. Principles and Techniques of Electron Microscopy, London, Macmillan, 1989, p288
- [Background] Barker AL, Konopatskaya O, Neal CR, Macpherson JV, Whatmore JL, Winlove CP, Unwin PR, Shore AC. Observation and characterisation of the glycocalyx of viable human endothelial cells using confocal laser scanning microscopy. Phys Chem Chem Phys 2004;6:1006-1011.
- [Background] van Zandvoort M, Engels W, Douma K, Beckers L, Oude Egbrink M, Daemen M, Slaaf DW. Two-photon microscopy for imaging of the (atherosclerotic) vascular wall: a proof of concept study. J Vasc Res. 2004 Jan-Feb;41(1):54-63. doi: 10.1159/000076246. Epub 2004 Jan 16. PMID 14730202
- [Background] Claesson-Welsh L. VEGF receptor signal transduction - A brief update. Vascul Pharmacol. 2016 Nov;86:14-17. doi: 10.1016/j.vph.2016.05.011. Epub 2016 Jun 4. PMID 27268035
- [Background] Olsson AK, Dimberg A, Kreuger J, Claesson-Welsh L. VEGF receptor signalling - in control of vascular function. Nat Rev Mol Cell Biol. 2006 May;7(5):359-71. doi: 10.1038/nrm1911. PMID 16633338
- [Background] Holmes K, Roberts OL, Thomas AM, Cross MJ. Vascular endothelial growth factor receptor-2: structure, function, intracellular signalling and therapeutic inhibition. Cell Signal. 2007 Oct;19(10):2003-12. doi: 10.1016/j.cellsig.2007.05.013. Epub 2007 Jun 12. PMID 17658244
- [Background] Pavlakovic H, Becker J, Albuquerque R, Wilting J, Ambati J. Soluble VEGFR-2: an antilymphangiogenic variant of VEGF receptors. Ann N Y Acad Sci. 2010 Oct;1207 Suppl 1(Suppl 1):E7-15. doi: 10.1111/j.1749-6632.2010.05714.x. PMID 20961309
- [Background] Stolz DB, Sims-Lucas S. Unwrapping the origins and roles of the renal endothelium. Pediatr Nephrol. 2015 Jun;30(6):865-72. doi: 10.1007/s00467-014-2798-3. Epub 2014 Mar 15. PMID 24633402
- [Background] Fu J, Lee K, Chuang PY, Liu Z, He JC. Glomerular endothelial cell injury and cross talk in diabetic kidney disease. Am J Physiol Renal Physiol. 2015 Feb 15;308(4):F287-97. doi: 10.1152/ajprenal.00533.2014. Epub 2014 Nov 19. PMID 25411387
- [Background] Munaut C, Lorquet S, Pequeux C, Coulon C, Le Goarant J, Chantraine F, Noel A, Goffin F, Tsatsaris V, Subtil D, Foidart JM. Differential expression of Vegfr-2 and its soluble form in preeclampsia. PLoS One. 2012;7(3):e33475. doi: 10.1371/journal.pone.0033475. Epub 2012 Mar 12. PMID 22428059
- [Background] van de Weg CA, Pannuti CS, van den Ham HJ, de Araujo ES, Boas LS, Felix AC, Carvalho KI, Levi JE, Romano CM, Centrone CC, Rodrigues CL, Luna E, van Gorp EC, Osterhaus AD, Kallas EG, Martina BE. Serum angiopoietin-2 and soluble VEGF receptor 2 are surrogate markers for plasma leakage in patients with acute dengue virus infection. J Clin Virol. 2014 Aug;60(4):328-35. doi: 10.1016/j.jcv.2014.05.001. Epub 2014 May 13. PMID 24928471
- [Background] Bonventre JV, Yang L. Cellular pathophysiology of ischemic acute kidney injury. J Clin Invest. 2011 Nov;121(11):4210-21. doi: 10.1172/JCI45161. Epub 2011 Nov 1. PMID 22045571
- [Background] Martensson J, Martling CR, Bell M. Novel biomarkers of acute kidney injury and failure: clinical applicability. Br J Anaesth. 2012 Dec;109(6):843-50. doi: 10.1093/bja/aes357. Epub 2012 Oct 9. PMID 23048068
- [Background] Kumar S, Liu J, McMahon AP. Defining the acute kidney injury and repair transcriptome. Semin Nephrol. 2014 Jul;34(4):404-17. doi: 10.1016/j.semnephrol.2014.06.007. Epub 2014 Jun 13. PMID 25217269
- [Background] Vaidya VS, Ozer JS, Dieterle F, Collings FB, Ramirez V, Troth S, Muniappa N, Thudium D, Gerhold D, Holder DJ, Bobadilla NA, Marrer E, Perentes E, Cordier A, Vonderscher J, Maurer G, Goering PL, Sistare FD, Bonventre JV. Kidney injury molecule-1 outperforms traditional biomarkers of kidney injury in preclinical biomarker qualification studies. Nat Biotechnol. 2010 May;28(5):478-85. doi: 10.1038/nbt.1623. PMID 20458318
- [Background] McIlroy DR, Wagener G, Lee HT. Biomarkers of acute kidney injury: an evolving domain. Anesthesiology. 2010 Apr;112(4):998-1004. doi: 10.1097/ALN.0b013e3181cded3f. No abstract available. PMID 20216399
- [Background] Kyoung KH, Hong SK. The duration of intra-abdominal hypertension strongly predicts outcomes for the critically ill surgical patients: a prospective observational study. World J Emerg Surg. 2015 May 30;10:22. doi: 10.1186/s13017-015-0016-7. eCollection 2015. PMID 26056530
- [Background] Herdan RA, Ibrahim AS, El-Gammal SAM, Bakr MAM, Latif MA, Ibraheem HA. Gastric Mucosal End-Tidal Carbon Dioxide Partial Pressure Difference as a Continuous Indicator of Splanchnic Perfusion During Prolonged Anesthesia. Med J Cairo Univ 2013; 18:(1): 359-65.
- [Background] Shokeir AA, Abubieh EA, Dawaba M, el-Azab M. Resistive index of the solitary kidney: a clinical study of normal values. J Urol. 2003 Aug;170(2 Pt 1):377-9. doi: 10.1097/01.ju.0000076620.27510.c4. PMID 12853779
- [Background] Antonetti DA, Barber AJ, Hollinger LA, Wolpert EB, Gardner TW. Vascular endothelial growth factor induces rapid phosphorylation of tight junction proteins occludin and zonula occluden 1. A potential mechanism for vascular permeability in diabetic retinopathy and tumors. J Biol Chem. 1999 Aug 13;274(33):23463-7. doi: 10.1074/jbc.274.33.23463. PMID 10438525
- [Background] Mehta D, Malik AB. Signaling mechanisms regulating endothelial permeability. Physiol Rev. 2006 Jan;86(1):279-367. doi: 10.1152/physrev.00012.2005. PMID 16371600
- [Background] Agarwal SK, Sethi S, Dinda AK. Basics of kidney biopsy: A nephrologist's perspective. Indian J Nephrol. 2013 Jul;23(4):243-52. doi: 10.4103/0971-4065.114462. PMID 23960337
- [Background] Schwarz A, Gwinner W, Hiss M, Radermacher J, Mengel M, Haller H. Safety and adequacy of renal transplant protocol biopsies. Am J Transplant. 2005 Aug;5(8):1992-6. doi: 10.1111/j.1600-6143.2005.00988.x. PMID 15996250
- [Background] Mostafa G, Greene FL. Fluid Management and Renal Function During a Laparoscopic Case Done Under CO2 Pneumoperitoneum. In: Scott-Conner CEH, editors. Fundamental of laparoscopy, thoracoscopy and GI Endoscopy. 2nd ed. New York: Springer; 2014.